CLINICAL TRIAL: NCT01834703
Title: Randomized Controlled Trial of Uterine Artery Embolization (UAE) Versus High-Intensity-Focused-Ultrasound (HIFU) for Treatment of Patients With Uterine Fibroids
Brief Title: Uterine Artery Embolization(UAE) Versus High-Intensity-Focused-Ultrasound(HIFU) for Treatment of Uterine Fibroids
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Simon Yu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIR-13-02
Record Dates: First submitted 2013-04-04; First posted 2013-04-18 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2016-02

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UAE treatment (Active Comparator): After randomization, patient recruited will be arranged to receive UAE treatment. 100 patients will be recruited for UAE treatment
  Interventions: Procedure: UAE
- HIFU (Active Comparator): After randomization, patient recruited will be arranged to receive HIFU treatment. 100 patients will be recruited for HIFU treatment
  Interventions: Procedure: HIFU

INTERVENTIONS:
Procedure: UAE — The patient will be admitted into hospital for UAE. UAE was performed with patients under local anesthesia. Embosphere particles (BioSphere Medical) with a size of 500 - 700µm were used in all procedures. Embospheres were mixed with contrast material and saline and injected into each uterine artery until either parenchyma filling of the fibroids had stopped (target embolization) or the main uterine artery was blocked with stasis of contrast material (selective embolization). After the procedure, women were admitted to the gynecology ward for postprocedural care. All patients were advised to stay in the hospital for at least 1 night.
  Arms: UAE treatment
Procedure: HIFU — Treatment will be given to the patient in one or more sessions on an outpatient basis. The uterine fibroid will be identified and located with ultrasonography and ablated with HIFU. For lesion beyond 6 cm distance from skin, HIFU is given at a power of 1200-1500 watt for 1500 - 2000 times at each spot, for 50 milli-second each time, at an interval of 100 milli-second, at a spot distance of 1.5cm, a line distance of 1.5cm, and a plane distance of 1.0 -1.5cm; for lesion within 6 cm distance from skin, HIFU is given at a power of 1300±15% Watt for 40 times at each spot, for120 milli-second each time, at an interval of 100 milli-second, at a spot distance of 0.3cm, a line distance of 0.3cm, and a plane distance of 0.8cm.
  Arms: HIFU

SUMMARY:
This study aimed to evaluate the clinical effectiveness and adverse effects of Uterine Artery Embolization (UAE), High-Intensity-Focused-Ultrasound (HIFU) in treating patients with uterine fibroid.

DETAILED DESCRIPTION:
The usual management for symptomatic uterine fibroid is surgery (myomectomy or hysterectomy), in the current study, uterine artery embolization (UAE) is a form of non-surgical and minimally invasive treatment, High-Intensity-Focused-Ultrasound (HIFU) is a form of non-invasive treatment that can be completed as an out-patient within hours. Embolization causes ischaemia and shrinkage of the fibroid and therefore symptomatic relieve. HIFU is a medical technology that has been used for cancer treatment. Energy is delivered from outside the body in a non-invasive manner to produce heat energy that causes necrosis and shrinkage of the uterine fibroid thereby relieves the symptoms due to the fibroid. It does not involve radiation. The clinical effectiveness of HIFU for uterine fibroid is unknown, however, based on the knowledge of the clinical effectiveness of HIFU on liver cancer and pancreatic cancer, there is reasonable ground to believe that HIFU is effective for uterine fibroid.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age between 30 and 47
* Pre or peri menopausal with Follicle-stimulating hormone (FSH) less than 40 mIU/ml
* Weight less than 140kg (or 310lbs) and Body Mass Index (BMI) less than 33
* Cervical cytology no more severe than low grade SIL
* Negative urine pregnancy test
* Uterine size less than 24 weeks based on physical exam assessment
* History of uterine leiomyoma causing symptoms of bleeding, pressure, or pain. Excessive uterine bleeding will be evidenced by either one of the following-profuse bleeding with flooding or clots or repetitive periods lasting for more than 8 days; or anemia due to acute or chronic blood loss OR pelvic discomfort caused by leiomyomata, either acute and severe or chronic lower abdominal or low back pressure or bladder pressure with urinary frequency not due to urinary tract infection
* Dominant intramural fibroid greater than or equal to 3 cm and less than or equal to 12 cm on imaging.
* Good health other than history of leiomyomas. Chronic medications may be acceptable at the discretion of the research team.
* No future fertility wish.
* Are using abstinence, mechanical (condoms, diaphragms) or sterilization methods of contraception and are willing to continue using them throughout the study.
* Willing and able to give informed consent.
* Willing and able to comply with study requirements.
* Normal menstrual cycle with endometrial pathology excluded
* Normal renal function
* Normal liver function
* Platelet count greater than 50 K/microL
* Normal coagulation profile

Exclusion Criteria:

* Significant abnormalities in the history, physical or laboratory examination
* History of or current thromboembolic event (deep vein thrombosis, pulmonary embolus, stroke)
* Other pelvic mass indicated by history or MR imaging such as endometriosis, ovarian tumor, acute or chronic pelvic inflammatory disease
* Desire for future pregnancy
* Pregnant or Positive pregnancy test
* Lactation
* Unexplained vaginal bleeding
* Untreated severe cervical dysplasia
* Intrauterine device
* Need for interval use of narcotics
* Extensive scarring along anterior lower abdominal wall (greater than 50% of area) or scar tissue or surgical clips in the direct path of the HIFU
* Pedunculated submucosal or subserosal fibroid of size ≧5cm and with a stalk less than 25% of the maximal fibroid diameter.
* Genetic causes of leiomyomata
* Known recent rapid growth of fibroids, defined as a doubling in size in 6 months
* Patient unwilling to receive non-surgical treatment
* Contraindication to MRI due to severe claustrophobia or implanted metallic device.

Ages: 30 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2009-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Treatment success rate | 6 months
  Technical success of treatment procedure and absence of symptoms of fibroid

SECONDARY OUTCOMES:
Incidence of procedure related complication | 1, 3, 6, 12 months after treatment
  Complications after treatment procedures will be recorded during each hospital admission and during each HIFU treatment session. Major adverse events will be reported. Complications that occur prior to a clinical visit will be documented and graded in each clinical visit at 1, 3, 6 and 12 month after treatment.
volume change of the fibroids | 6, 12 months after treatment
  Assessed by 3 Dimensional ultrasonography (USG)
Degree of infarction of the fibroids | 3, 15 months after treatment
  Contrast enhanced magnetic resonance imaging (MRI) is used to assess the degree of infarction, which is defined as non-perfused tissue on contrast MRI.
Vascularity of the fibroids | 6, 12 months after treatment
  Assessed by contrast enhanced USG. Vascularity of the fibroid will be classified into six categories: 0%, <25%, 25 to 50%, >50 to 75%, >75%, 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Simon CH Yu, MD, FRCR, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Department of Imaging and Interventional Radiology, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong
  - Department of Obstectrics and Gynaecology, Prince of Wales Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No